CLINICAL TRIAL: NCT05938491
Title: OCT and OCT Angiography After Diabetic Vitrectomy With or Without Internal Limiting Membrane Peeling for Patients With PDR
Brief Title: OCT and OCT-A Afer Diabetic Vitrectomy in PDR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Abdelkarem Hasan, Assistant lecturer of ophthalmology, Assiut University
Other Study IDs: oct after diabetic vitrectomy
Record Dates: First submitted 2023-06-26; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: OCT and OCT-A — OCT and OCT angiography for the macula

SUMMARY:
Detection of any structural or vascular changes at the macula after Pars Plana Vitrectomy ( PPV ) in cases with complicated proliferative diabetic retinopathy ( PDR )

ELIGIBILITY:
Inclusion Criteria:

* Cases with complicated PDR as persistant vitreous hemorrhage or tractional retinal detachment involving or threatening the macula underwent PPV with or without ILM peeling

Exclusion Criteria:

* eyes with media opacity after PPV not allowing imaging of the macula

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with complicated proliferative diabetic retinopathy underwent pars plana vitrectomy
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
OCT and OCT angiography to assess the macular thickness , outline and vascularity | 3 months after surgery
  Detection of any structural or vascular changes at the macula after Pars Plana Vitrectomy ( PPV ) in cases with complicated proliferative diabetic retinopathy ( PDR ) .

IPD SHARING:
Plan to Share IPD: Undecided